CLINICAL TRIAL: NCT01264601
Title: Multi-Centered, Randomized, Placebo-Controlled Trial of the Safety of Influenza Vaccine in Egg Allergic Children With a History of Anaphylaxis or Severe Allergy to Egg
Brief Title: Safe Administration of Flu Vaccine to Egg Allergic Children
Acronym: SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American College of Allergy, Asthma and Immunology (Other)
Responsible Party: Principal Investigator, Matthew Greenhawt, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM 00038826
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Results first posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Egg Allergy
Keywords: Anaphylaxis to Egg; Severe Egg Allergy
MeSH Terms: conditions — Egg Hypersensitivity | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single Dose (Experimental): This arm will receive TIV as 2 doses, the first of which will be normal saline administered at approximately 10% of the total age appropriate dose volume, followed 30 minutes later by the full age appropriate dose. For children receiving a 0.25ml dose, a 20%/80% split will be used for ease of administration in drawing up the dose.
  Interventions: Biological: Trivalent Influenza Vaccine
- Graded Challenge (Experimental): Subjects in this arm will receive TIV by standard 10%/90% 2-step graded challenge split of the age appropriate dose, separated by 30 minutes. For children receiving a 0.25ml dose, a 20%/80% split will be used for ease of administration in drawing up the dose.
  Interventions: Biological: Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: Trivalent Influenza Vaccine — Age appropriate dose of seasonal Trivalent Influenza Vaccine (TIV), either 0.25mL under age 3 or 0.5mL over the age of 3.

SUMMARY:
Historically, providing influenza vaccination of egg allergic children and young adults (EAC) with a history of anaphylaxis to egg, or other severe symptoms of an allergic reaction to egg (e.g., severe hives, swelling, or asthma), has been contra-indicated, though vaccination of children with less severe egg allergy has been shown to be safe. Though many children with severe egg allergy, including anaphylaxis, have received past influenza vaccination anecdotally, very few data exist to show this procedure is safe. The investigators propose a double blind, placebo-controlled randomized, prospective multi-centered study to a) demonstrate seasonal trivalent influenza vaccine (TIV) can be safely given in a single dose (as opposed to through 2-step graded dosing of 10% then 90% of the vaccine dose) to EAC despite history of anaphylaxis or previous severe allergic reaction to egg; and b) provide further evidence that adverse outcomes are not related to ovalbumin (egg) content in TIV.

Study participants must have a documented history of a severe egg allergy, substantiated by both a history of clinical reactivity AND either a positive skin test or ImmunoCAP/RAST test greater than 0.7 kUA/L. Participants will be randomized to receive either a 2-step graded challenge or a single dose given after a small placebo dose of saline (to mimic the graded challenge). If required, all participants will receive a booster vaccination as a single dose.

DETAILED DESCRIPTION:
Seasonal Trivalent Influenza Vaccine (TIV) is grown in embryonated chicken eggs, and since it contains residual egg protein (ovalbumin), providing TIV to egg allergic children (EAC) could potentially provoke allergic reactivity. Because of this possibility, historically caution has been advised in providing TIV to these children, and the vaccine has been withheld in certain individuals, though for many it has been safely administered after vaccine skin testing and stepwise administration. In the 2009 American Academy of Pediatrics Red Book (and previous editions), a history of severe allergic reactivity to egg is a contraindication to receiving TIV, though it is acknowledged that less severely egg allergic kids have safely received TIV if precautions had been taken.

In the past year, several studies have emerged that demonstrate that most, if not all, EAC can safely be vaccinated with both TIV ad the H1N1 vaccine. A recent 5 year review of TIV administration in EAC ages 6 mo-36 mo, showed safe administration to 135 EAC after TIV skin testing, including 14 subjects with a history of anaphylaxis to egg. Another large, retrospective study of non-anaphylactic EAC showed TIV could be successfully administered using a 2-step protocol without skin testing to TIV. In a single center H1N1 vaccine study last fall, 105 EAC received either a full vaccine dose if skin tests were negative, or a 2-step graded challenge if the tests were positive, including 25 subjects with a history of anaphylaxis. No allergic reactions resulted, regardless of the results of skin testing, the method of administration, ovalbumin content of the vaccine, or use of a different booster lot without pre-testing. In a sister-study, 68 H1N1 participants prospectively received TIV safely without graded challenge, including 13 EAC with a history of egg anaphylaxis. A large prospective, Canadian multi-centered study, using an adjuvanted H1N1 preparation containing 0.03μg/mL of ovalbumin, was safely given to 72 individuals with either a history of severe cardiopulmonary reactivity to egg or a history of poorly controlled asthma (this group was not further broken down), via 2-step graded challenge. Thus, these studies suggest it is safe for EAC with a history of anaphylaxis to receive TIV and H1N1 without pre-testing, suggest that use of a 2-step graded challenge may be unnecessary, and show some evidence that past egg allergy severity may not be an important factor in vaccine tolerance. Recent guidelines published by the AAAAI suggest a flexible approach is reasonable, and that EAC can receive TIV without prior skin testing through either a single dose or a 2-step approach.

This double blind, randomized, placebo-controlled, multi-centered study aims to investigate the safety of TIV given to EAC with a history of a severe past reaction or anaphylaxis to egg, and aims to show that a single dose route of administration is safe and sufficient. Participants with new or established severe egg allergy (see eligibility criteria) will be randomized to receive either a 2-step (10%, followed by 30 min. observation, then residual 90%) graded challenge or a single dose of TIV given 30 minutes after a placebo dose of normal saline is administered (to approximate the graded challenge). Vaccine tolerance will be analyzed and compared to ovalbumin content of the vaccine lots, as well as to baseline characteristics of the participant's egg allergy and allergic history.

Secondary outcomes originally posted on the www.clinicaltrials.gov website were hypotheses which were aims of complex data analysis but were not in and of themselves actual outcome measures. Therefore these have been deleted from the record

ELIGIBILITY:
Inclusion Criteria:

1. Ages 6 months-24 years, seen in the UMHS Allergy Clinics (and similar academic Allergy clinics of collaborating sites) in the last 24 months with a discharge diagnosis code of v15.03 indicating an of egg allergy, AND with correlated history including the following:

   1. Egg allergy as defined by:

      Positive egg challenge; OR strong history suggestive of clinical allergy within 4 hours of ingestion AND egg-specific IgE above 0.70 kUA/L OR wheal 3mm > control (or 2+ score if wheal size not available).
   2. Anaphylaxis after egg ingestion, defined by:

   Patients with a verified history (by chart review) of their single most severe reaction to egg resulting in the following, per NIAID/FAAN 2006 criteria:5 i) Acute onset of an illness with involvement of the skin/mucosal tissue (e.g., generalized hives, pruritus or flushing, swollen lips-tongue-uvula) AND EITHER respiratory compromise (e.g., dyspnea, wheezing/bronchospasm, stridor, reduced peek expiratory flow) OR reduced blood pressure or associated symptoms (eg, hypotonia or syncope); OR ii) Two or more of the following after exposure to an allergen: involvement of the skin/mucosal tissue (e.g., urticaria, itching/flushing, swollen lips/tongue/uvula); respiratory compromise (e.g., dyspnea, wheezing/bronchospasm, stridor, reduced peak expiratory flow); reduced blood pressure or associated symptoms (e.g., hypotonia or syncope); or persistent gastrointestinal symptoms (e.g., crampy abdominal pain or vomiting); OR iii) Hypotension after exposure to known allergen for that patient c) A severe allergic reaction will be defined by a history of development of severe hives, angioedema, or allergic asthma attributable to egg allergy.
2. Subject must fulfill criteria for both egg allergy and for either anaphylaxis or a severe allergic reaction (both attributable to egg) to be included in the study, i.e. both (a) and either (b) or (c).
3. Ability to remain off antihistamines for at least 5 days prior to the study visit, for skin testing.
4. For children, the ability to remain in the exam room for the duration of the testing visit.
5. Previous history of TIV of H1N1 vaccination is neither inclusive nor exclusive for the study.

Exclusion Criteria:

1. Does not fulfill requirements for both egg allergy AND anaphylaxis or severe allergic reaction.
2. Prolonged use of immunosuppressive medication, including high dose corticosteroids > 6 months, as well as other immunosuppressive agents.
3. Prior history of egg allergy, now outgrown and tolerating egg ingestion.
4. Eosinophilic esophagitis.
5. Cardiac disease.
6. Known malignancy under treatment.
7. Pregnant women.

Ages: 6 Months to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Greenhawt, MD, MBA, Principal Investigator — University of Michigan; Georgiana Sanders, MD, MS, Principal Investigator — University of Michigan
Locations (5):
- United States (5):
  - Scripps Clinic, San Diego, California
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Children's Hospital of Pittsburgh, University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, University of Texas-Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Background] American Academy of Pediatrics. Influenza. In: Pickering LK, ed. Red Book: 2009 Report of the Committee on Infectious Diseases. 28th ed. Elk Grove Village, IL: American Academy of Pediatrics; 2009:400-412. Available at: http://aapredbook.aappublications.org/cgi/content/full/2009/1/3.64. Accessed June 18, 2010.
- [Background] Howe LE, Chernin A, Sanders GM. Administration of Influenza Vaccine to the Egg Allergic Child Under 36 Months (Abstract). J Allergy Clin Immunol 2010; 125:AB23.
- [Background] Greenhawt MJ, Chernin AS, Howe L, Li JT, Sanders G. The safety of the H1N1 influenza A vaccine in egg allergic individuals. Ann Allergy Asthma Immunol. 2010 Nov;105(5):387-93. doi: 10.1016/j.anai.2010.08.015. PMID 21055666
- [Background] Gagnon R, Primeau MN, Des Roches A, Lemire C, Kagan R, Carr S, Ouakki M, Benoit M, De Serres G; PHAC-CIHR Influenza Research Network. Safe vaccination of patients with egg allergy with an adjuvanted pandemic H1N1 vaccine. J Allergy Clin Immunol. 2010 Aug;126(2):317-23. doi: 10.1016/j.jaci.2010.05.037. Epub 2010 Jun 25. PMID 20579720
- [Background] Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol. 2006 Feb;117(2):391-7. doi: 10.1016/j.jaci.2005.12.1303. PMID 16461139
- [Background] Chung EY, Huang L, Schneider L. Safety of influenza vaccine administration in egg-allergic patients. Pediatrics. 2010 May;125(5):e1024-30. doi: 10.1542/peds.2009-2512. Epub 2010 Apr 5. PMID 20368312
- [Background] Li JT, Rank MA, Squillace DL, Kita H. Ovalbumin content of influenza vaccines. J Allergy Clin Immunol. 2010 Jun;125(6):1412-3; author reply 1413-4. doi: 10.1016/j.jaci.2010.03.009. Epub 2010 May 7. No abstract available. PMID 20451987
- [Background] Waibel KH, Gomez R. Ovalbumin content in 2009 to 2010 seasonal and H1N1 monovalent influenza vaccines. J Allergy Clin Immunol. 2010 Mar;125(3):749-51, 751.e1. doi: 10.1016/j.jaci.2009.12.015. Epub 2010 Jan 8. No abstract available. PMID 20060576
- [Background] James JM, Zeiger RS, Lester MR, Fasano MB, Gern JE, Mansfield LE, Schwartz HJ, Sampson HA, Windom HH, Machtinger SB, Lensing S. Safe administration of influenza vaccine to patients with egg allergy. J Pediatr. 1998 Nov;133(5):624-8. doi: 10.1016/s0022-3476(98)70101-5. PMID 9821418
- [Background] Zeiger RS. Current issues with influenza vaccination in egg allergy. J Allergy Clin Immunol. 2002 Dec;110(6):834-40. doi: 10.1067/mai.2002.129372. PMID 12464947
- [Background] Kelso JM. Administration of influenza vaccines to patients with egg allergy. J Allergy Clin Immunol. 2010 Apr;125(4):800-2. doi: 10.1016/j.jaci.2010.02.013. Epub 2010 Mar 11. No abstract available. PMID 20226505
- [Background] Greenhawt MJ, Li JT, Bernstein DI, Blessing-Moore J, Cox L, Khan D, Lang DM, Nicklas RA, Oppenheimer J, Portnoy JM, Randolph C, Schuller DE, Spector SL, Tilles SA, Wallace D. Administering influenza vaccine to egg allergic recipients: a focused practice parameter update. Ann Allergy Asthma Immunol. 2011 Jan;106(1):11-6. doi: 10.1016/j.anai.2010.11.015. No abstract available. PMID 21195939
- [Background] Webb L, Petersen M, Boden S, LaBelle V, Bird JA, Howell D, Burks AW, Laubach S. Single-dose influenza vaccination of patients with egg allergy in a multicenter study. J Allergy Clin Immunol. 2011 Jul;128(1):218-9. doi: 10.1016/j.jaci.2011.02.013. Epub 2011 Apr 2. No abstract available. PMID 21459425

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from October 2010 through March 2012 at the University of Michigan.
Pre-assignment Details: After informed consent process, parents filled out a questionnaire, detailing their child's history of past reactions to the ingestion of egg and any prior influenza vaccines. This information was verified by medical record review. In addition, the most recent egg skin test and serum egg protein specific IgE were also obtained.
Groups:
- Single Dose: This arm will receive TIV as 2 doses, the first of which will be normal saline administered at approximately 10% of the total age appropriate dose volume, followed 30 minutes later by the full age appropriate dose. For children receiving a 0.25ml dose, a 20%/80% split will be used for ease of administration in drawing up the dose.
  Trivalent Influenza Vaccine : Age appropriate dose of seasonal Trivalent Influenza Vaccine (TIV), either 0.25mL under age 3 or 0.5mL over the age of 3.
- Graded Challenge: Subjects in this arm will receive TIV by standard 10%/90% 2-step graded challenge split of the age appropriate dose, separated by 30 minutes. For children receiving a 0.25ml dose, a 20%/80% split will be used for ease of administration in drawing up the dose.
  Trivalent Influenza Vaccine : Age appropriate dose of seasonal Trivalent Influenza Vaccine (TIV), either 0.25mL under age 3 or 0.5mL over the age of 3.
Period: Overall Study
Arm/Group | Single Dose | Graded Challenge
Started | 17 | 14
Completed | 17 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose | Graded Challenge | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 14 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.6 (3.4) | 6.3 (5.1) | 6.2 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 10 | 6 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 14 | 31
Egg skin test wheal, median, mm [Median (Standard Deviation); unit: mm] | 9 (3.4) | 6 (4.2) | 7 (3.5)
Prior TIV [Count of Participants; unit: Participants] | 12 | 11 | 23
Prior H1N1 Vaccine [Count of Participants; unit: Participants] | 10 | 6 | 16
History of Anaphylaxis to Egg [Count of Participants; unit: Participants] | 8 | 6 | 14
Baked Egg Tolerant [Count of Participants; unit: Participants] | 5 | 5 | 10
Atopic Dermatitis [Count of Participants; unit: Participants] | 8 | 10 | 18
Asthma [Count of Participants; unit: Participants] | 7 | 4 | 11
Allergic Rhinitis [Count of Participants; unit: Participants] | 3 | 5 | 8
Other Food Allergy [Count of Participants; unit: Participants] | 12 | 7 | 19
Serum Specific IgE Egg White [Median (Standard Deviation); unit: Measured in kUA/L] | 5.3 (23.6) | 16.2 (28.9) | 10.2 (25)
Serum Specific IgE Ovalbumin [Median (Standard Deviation); unit: kUA/L] | 4.52 (25.2) | 10.45 (35.5) | 7.1 (25.2)
Serum Specific IgE Ovomucoid [Median (Standard Deviation); unit: kUA/L] | 2.83 (28) | 7 (39.8) | 4.32 (24.4)
Localized Urticaria [Count of Participants; unit: Participants] | 6 | 5 | 11
Systemic Urticaria [Count of Participants; unit: Participants] | 9 | 5 | 14
Oral/Facial Angioedema [Count of Participants; unit: Participants] | 5 | 6 | 11
Throat Itching [Count of Participants; unit: Participants] | 3 | 3 | 6
Throat Swelling [Count of Participants; unit: Participants] | 1 | 2 | 3
Stridor [Count of Participants; unit: Participants] | 2 | 1 | 3
Cough [Count of Participants; unit: Participants] | 10 | 3 | 13
Dyspnea [Count of Participants; unit: Participants] | 1 | 2 | 3
Wheezing [Count of Participants; unit: Participants] | 2 | 2 | 4
Hypotension [Count of Participants; unit: Participants] | 1 | 1 | 2
Vomiting [Count of Participants; unit: Participants] | 10 | 9 | 19
Abdominal Pain [Count of Participants; unit: Participants] | 2 | 3 | 5
Age at Diagnosis [Median (Standard Deviation); unit: months] | 12 (19.5) | 11 (14.4) | 12 (17.6)

OUTCOME MEASURES:

1. Primary Outcome: Categorical Reactivity to Vaccine as it Was Administered
Description: After randomization, group 1 will receive a 10%/90% (or 20%/80% for 0.25ml) graded challenge of the age appropriate TIV dose, separated by 30 minutes for observation. Group 2 will receive a first dose consisting of normal saline at a volume equal to 10% of their age appropriate dose, and the second dose will consist of their full age appropriate dose as the "90%" equivalent, also separated by 30 minutes of observation. For children receiving a 0.25ml dose, a 20%/80% split will be used for ease of administration in drawing up the dose. All parties will report any adverse reactions occurring in the next 48 hours after vaccination that were not observed at the time of in office observation.
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose | Graded Challenge
Number analyzed (Participants) | 17 | 14
Participants
  No systemic reactivity | 17 | 14
  Mild, transient, induration at injection site | 3 | 4

2. Secondary Outcome: Influence of Atopic Co-morbidities on Severe Reactivity to Vaccine as it Was Administered
Description: Rates of co-morbid allergic disease, size and magnitude of egg skin and ImmunoCAP tests, presence of other food allergy, and tolerance of "baked egg" will be assessed through a screening questionnaire and chart review, and compared between the groups to assess for any significant differences that may predict TIV tolerance.
Time Frame: 6 months
Population: Because no participants had systemic/severe reactivity, there were no participants who were TIV intolerant, and therefore no meaningful analysis of correlation of baseline characteristics to intolerance could be performed. All Baseline Characteristics collected for the original purpose of such correlation are reported in Baseline Characteristics.
Arm/Group | Single Dose | Graded Challenge
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Single Dose | Graded Challenge
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 1/17 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose (N=17) | Graded Challenge (N=14)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — 2 year old boy vomited app. 28 min. post-vaccination after vigorously running around. Was otherwise playful and no other symptoms of IgE-mediated reactivity. Per the PIs at Univ. of Michigan, this event was believed to be unrelated to the study.
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — 12 yr old boy, receiving first TIV, reported Tachycardia 24 hours after vaccincation but no symptoms noted during observation period or later on same day/night. Per the PIs at the Univ. of Michigan, event believed to be unrelated to the study.
Anaphylaxis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — A 3 yr old with milk and egg allergy developed anaphylaxis within few min. of consuming a chocolate sauce labeled as having both milk and egg, app. 24 hours after vaccine. Per the PIs at Univ. of Mich., this event believed unrelated to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes